CLINICAL TRIAL: NCT06315244
Title: Effectiveness of Perforating Cutaneous Nerve Injection in Patients With Chronic Coccydynia: A Prospective, Randomized, Placebo-Controlled, Double-Blind Study
Brief Title: Perforating Cutaneous Nerve Injection Efficacy in Chronic Coccydynia: A Randomized, Double-Blind Study
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Enes Efe Is, MD, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2558
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Coccyx Disorder; Coccyx Injury

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- %5 Dextrose Injection Group (Experimental): Participants in this arm will receive an ultrasound-guided injection of 5% dextrose solution into the sacrotuberous ligament and the sensory innervation area of the perforating cutaneous nerve. The intervention aims to alleviate symptoms of chronic coccydynia by reducing nerve entrapment. Participants will continue their existing physical therapy/medical treatment regimen throughout the study.
  Interventions: Procedure: US Guided Perineural Injection and Neuroprolotherapy
- Placebo Injection Group (Placebo Comparator): Participants in this arm will receive an ultrasound-guided injection of a placebo solution (saline) into the same anatomical region as the experimental group. This arm serves as a control to evaluate the efficacy of the dextrose injection in treating chronic coccydynia symptoms. Participants will continue their existing physical therapy/medical treatment regimen throughout the study.
  Interventions: Procedure: US Guided Perineural Injection and Neuroprolotherapy

INTERVENTIONS:
Procedure: US Guided Perineural Injection and Neuroprolotherapy — Participants will receive an ultrasound-guided injection of a solution into the sacrotuberous ligament and the sensory innervation area of the perforating cutaneous nerve.

SUMMARY:
Interventions targeting the perforating cutaneous nerve are relatively new to the literature, with a safe side-effect profile but lacking high-quality studies. Their effectiveness remains at the level of case presentations. According to the hypothesis expressed in these publications, coccydynia might be an overlooked cause due to the compression of the perforating cutaneous nerve where it pierces the sacrotuberous ligament and becomes superficial. Ultimately, it is hypothesized that injection of dextrose into this ligament and the sensory area of this nerve will resolve these symptoms due to nerve entrapment, similar to other entrapment neuropathies treated with 5% dextrose, like carpal tunnel syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 50 years.
2. Chronic coccyx pain (≥3 months).
3. Pain Visual Analogue Scale (VAS) score ≥4.
4. Pain not alleviated by first-line treatment (physical therapy/oral analgesic therapy + sitting cushion).

Exclusion Criteria:

1. Injection to the area in the last 3 months.
2. Concurrent mechanical or inflammatory low back pain.
3. Coccyx pain that started during pregnancy or postpartum.
4. History of myelomeningocele or spina bifida.
5. History of sacrococcygeal luxation or subluxation (confirmed by radiography).
6. History of coccyx fracture.
7. Concurrent neurological deficit.
8. Skin disease affecting the injection area.
9. History of malignancy.
10. Pregnancy or breastfeeding.
11. Severe coagulopathy.
12. Infection at the injection site.
13. Neurological or psychiatric diseases, including ongoing depression (Beck Depression Inventory Score >14).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of Perforating Cutaneous Nerve Injection | Baseline, 2 weeks, 1 month, and 3 months post-treatment
  To evaluate the effectiveness of perforating cutaneous nerve injection in reducing pain in patients with chronic coccydynia. Pain levels will be assessed using the Visual Analogue Scale (VAS) during sitting, movement and rest.

SECONDARY OUTCOMES:
Change in Pressure Pain Threshold | Baseline, 2 weeks, 1 month, and 3 months post-treatment
  Assessment of the pressure pain threshold using an algometer.
Change in Quality of Life | Baseline, 2 weeks, 1 month, and 3 months post-treatment
  Assessment of quality of life using the EuroQoL questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Julide Oncu Alptekin, Professor, Study Chair — Sisli Hamidiye Training and Research Hospital
Locations (1):
- Sisli Hamidiye Etfal Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided